CLINICAL TRIAL: NCT00792974
Title: End-of-Life Fear in Patients With End-Stage Lung Disease: Fears of Death and Dying, Wishes and Needs of Patients With Severe COPD
Brief Title: End-of-Life Fear in Patients With End-Stage Lung Disease (COPD)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Philipps University Marburg (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Prof. Dr. W. Rief, Department of Clinical Psychology and Psychotherapy
Other Study IDs: EoL
Record Dates: First submitted 2008-11-17; First posted 2008-11-18 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; End-of-Life Fear; Fear About Death and Dying; Depression
Keywords: Cognitive behavioral education; COPD (Chronic Obstructive Pulmonary Disease), GOLD II-IV
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Depression | interventions — Cognitive Behavioral Therapy; Palliative Care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- COPD by GOLD-criteria III and IV
  Interventions: Behavioral: A brief psycho-educational intervention

INTERVENTIONS:
Behavioral: A brief psycho-educational intervention — A brief (3 single sessions) psycho-educational program with cognitive-behavioral and disease self-management techniques.
  This study is an open pilot study ("feasibility study") to develop a palliative psychological program for end-of-life fears in COPD, therefore all participants will be given the opportunity to receive treatment.
  Other Names: Cognitive-behavioral therapy; Palliative care

SUMMARY:
The aim of the study is to develop an interview to ask patients with COPD about their fear of death and dying, their needs and wishes at the end-of-life. Afterwards, the patients receive a brief psychological intervention to develop coping strategies for chronic illness. Beside this a general purpose of this intervention is to improve patients' quality of life.

DETAILED DESCRIPTION:
Background:

COPD-related mortality differs markedly from that of other chronic diseases. While the mortality rates for heart disease and stroke have fallen significantly, death rates caused by COPD have more than doubled. Therefore there is a major need to address questions of palliative end-of-life care. Patients with end-stage pulmonary lung diseases suffer from dyspnea, severe pain, fatigue and - the "deadlock" in end-of-life communication. Many people with severe COPD are socially isolated, have low quality of life and psychosocial challenges such as sadness, panic or hopelessness. In fact, 70 up to 90% suffer from a clinically relevant depression and/or anxiety disorder. Despite this, the majority of COPD patients with co-morbid disorders don't receive any treatment for their psychological symptoms. Furthermore, there is substantial evidence that only a minority of people with end-stage COPD have the opportunity to discuss their fears and wishes for end-of-life care. The few existing studies on this issue demonstrated that the majority of people with severe COPD wants to discuss topics such as prognosis, fear of death and dying or preferences and needs at the end-of-life. Understanding the nature and implications of treatment options is an important component of advanced care planning for people with end-stage lung disease.

Therefore the aim of this study is to bring up the end-of-life communication to patients with end-stage COPD. We hypothesize that end-stage COPD patients have greater fear of death and dying as patients with mild to moderate COPD or with hip prothesis (control group). The lowest anxiety rate with regard to death should be found in the healthy control group. Furthermore, a brief psychological intervention should decrease the co-morbid psychological symptoms and patients' fears. Higher quality of life should be achieved.

Objectives:

Subjects are recruited from the Pulmonary Rehabilitation Units of the Berchtesgadener Klinikum Schönau, Germany, through direct recruitment and use of administrative databases. All patients providing informed consent are invited to participate, if they have a chronic obstructive pulmonary disease with stage II, III or IV by GOLD-criteria. An open three group comparison is made of one-hundred patients with severe COPD (stage III and IV), thirty-three patients with moderate COPD (stage II), thirty-three patients with hip prosthesis and thirty-three mental healthy persons matched for age and sex. As we want to start a first feasibility intervention study, this is a clinical controlled design without randomization.

Methods:

Initially a systematic literature review was performed to determine what methods are being used in COPD studies and how the patients' views can be best assessed. Then a qualitative multi-method design will be used involving semi-structured interviews, standardized questionnaires and lung function parameters.

The face-to-face interview includes ten categories with more than 70 questions on

1. social demography
2. actual health status
3. knowledge and wishes of further information about the disease
4. thoughts and attitudes about the illness
5. fears about the illness, treatment and prognosis
6. general experiences of death and dying
7. own experiences with death and dying
8. fear of death
9. fear of dying
10. end-of-life decisions such as wishes and needs

Patients will be interviewed by a single interviewer. Each question will be read by using everyday language. Interviews will be audiotaped to control for integrity. Each interview will last approximately 60 minutes. The interview will be validated by the COPD-Anxiety-Questionnaire (CAF). To assess the patients cognitions about death, a self-report questionnaire, FIMEST, will be also used.

Standardized questionnaires will be used to detect depression or panic disorders by the Hospital Anxiety and Depression Scale. Functional health status will be measured by the Patients Health Questionnaire (PHQ) and the COPD-Disability- Index (CDI). The condition specific questionnaire, the Short Form-36 Health Survey (SF-36) and Euroqol (EQ) will be compared for their discriminative and evaluative properties. Spirometric tests and a walking test will be also performed.

After the interview those patients who have increased death anxiety take part in a brief psychological intervention to discuss their end-of-life issues, worries and fears. For this psychological intervention, a manualized 2-3-session approach will be used.

ELIGIBILITY:
Inclusion Criteria:

* 50 years or older
* COPD diagnosis III and IV by GOLD-criteria with or without an indication for long-term oxygen therapy (LTOT), non invasive ventilation (NIV) and/or lung transplantation (LTx)
* COPD diagnosis II by GOLD-criteria
* Patients with hip prosthesis
* Mental healthy people, who have no severe illness (such as heart disease or cancer) one year before

Exclusion Criteria:

* Participation in other studies likely to influence the patient in terms of confounding effects
* Acute and severe exacerbations with hard symptoms over 4 days
* Patients need a increasing medication of steroids and/or antibiotics
* Non-compliance

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects are recruited from the Pulmonary Rehabilitation Units of the Berchtesgadener Klinikum Schönau, Germany, through direct recruitment and use auf administrative databases. All patients who are alert and can provide consent are invited to participate, if they have a chronic obstructive pulmonary disease with stage II, III or IV by GOLD-criteria. An open three group comparison is made of one-hundred patients with severe COPD (stage III and IV), thirty-three patients with moderate COPD (stage II), thirty-three patients with hip prosthesis and thirty-three mental healthy persons in match-able age.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-07 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Self-reported semi-structured interview about the fear of death and dying, needs and wishes at the end-of-life in patients with severe COPD | Pre-Post-Design including 2 assessment points: pre-treatment and post-treatment

SECONDARY OUTCOMES:
St. George's Respiratory Questionnaire (SGRQ) | Pre-Post-Design including 2 assessment points: pre-treatment and post-treatment
Short Form Health Survey (Fragebogen zum allgemeinen Gesundheitszustand, SF-36) | Pre-Post-Design including 2 assessment points: pre-treatment and post-treatment
Euroqol (EQ) | Pre-Post-Design including 2 assessment points: pre-treatment and post-treatment
Patient Health Questionnaire (PHQ) | Pre-Post-Design including 2 assessment points: pre-treatment and post-treatment
Hospital Anxiety and Depression Scale (HADS) | Pre-Post-Design including 2 assessment points: pre-treatment and post-treatment
Borg Scale | Pre-Post-Design including 2 assessment points: pre-treatment and post-treatment
Diffusion capacity (DLCO) | Pre-Post-Design including 2 assessment points: pre-treatment and post-treatment
Blood gas analysis (BGA) | Pre-Post-Design including 2 assessment points: pre-treatment and post-treatment
Bodyplethysmographs | Pre-Post-Design including 2 assessment points: pre-treatment and post-treatment
Bio-Impedance-Analysis (BIA) | Pre-Post-Design including 2 assessment points: pre-treatment and post-treatment
6-Minute Walk Distance (6 MWD) | Pre-Post-Design including 2 assessment points: pre-treatment and post-treatment
Body Mass Index (BMI) | Pre-Post-Design including 2 assessment points: pre-treatment and post-treatment
Blood tests | Pre-Post-Design including 2 assessment points: pre-treatment and post-treatment
Multidimensional assessment of attitudes toward death and dying (Fragebogeninventar zur mehrdimensionalen Erfassung des Erlebens gegenüber Sterben und Tod, FIMEST) | Pre-Post-Design including 2 assessment points: pre-treatment and post-treatment
COPD- Anxiety -Questionnaire (COPD-Angst-Fragebogen, CAF) | Pre-Post-Design including 2 assessment points: pre-treatment and post-treatment
COPD- Disability- Index (CDI) | Pre-Post-Design including 2 assessment points: pre-treatment and post-treatment
Differences in COPD admission rates, functional impairment, quality of life and end-of-life fear after treatment | Pre-Post-Design including 2 assessment points: pre-treatment and post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Rief, Prof. Dr., Principal Investigator — Department of Clinical Psychology and Psychotherapy, Philipps University Marburg, Germany; Klaus Kenn, Dr., Study Director — Klinikum Berchtesgadener Land, Schön Kliniken, Schönau a. K., Germany; Sabine R Pinzer, Dipl.-Psych., Study Chair — Department of Clinical Psychology and Psychotherapy, Philipps University Marburg, Germany
Locations (2):
- Germany (2):
  - Department of Clinical Psychology and Psychotherapy, Philipps University Marburg, Marburg
  - Klinikum Berchtesgadener Land, Schön Kliniken, Schönau am Königssee